CLINICAL TRIAL: NCT01016808
Title: A Randomized, Double-Blind, Multi-Center, Repeat-Dose, Comparison of the Analgesic Efficacy and Safety of Q8003 With Oxycodone and Morphine for the Management of Acute Moderate to Severe Postoperative Pain Following Bunionectomy Surgery
Brief Title: Comparison of the Efficacy and Safety of Q8003 Versus Its Individual Components in Bunionectomy Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: QRxPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Q8003-008
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Moderate to Severe Postoperative Pain
Keywords: Bunionectomy; Opioids
MeSH Terms: interventions — MoxDuo; Morphine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Q8003 12 mg/8 mg (Experimental): Combination
  Interventions: Drug: Q8003
- Morphine sulfate 12 mg (Active Comparator): Single component
  Interventions: Drug: Morphine sulfate
- Oxycodone HCl 8 mg (Active Comparator): Single component
  Interventions: Drug: Oxycodone HCl

INTERVENTIONS:
Drug: Q8003 — Q8003 is a combination of morphine sulfate and oxycodone HCl
  Arms: Q8003 12 mg/8 mg
Drug: Morphine sulfate — One morphine sulfate 12 mg IR capsule q6h
  Arms: Morphine sulfate 12 mg
Drug: Oxycodone HCl — One oxycodone HCl 8 mg IR Capsule q6h
  Arms: Oxycodone HCl 8 mg

SUMMARY:
This is a randomized, double-blind, multicenter, fixed dose factorial study of Q8003 12 mg/8 mg versus its individual morphine sulfate and oxycodone hydrochloride components for the management of acute moderate to severe postoperative pain following bunionectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female and at least 18 years of age.
* Females must be non-pregnant, non-lactating, and practicing an acceptable method of birth control, or be surgically sterile or postmenopausal (amenorrhea for ≥ 12 months). Non-pregnancy will be confirmed by pregnancy tests conducted at Screening and Pre-treatment.
* Patient is scheduled for bunionectomy surgery, meets the criteria of an ASA Class I to III, and is willing to stay in the study center for at least 48 hours from the initial dose of study medication post surgery.
* To be randomized after surgery, the patient must report moderate to severe pain (a score of 2 or more on the 4 point Likert scale or at least 4 on the 11 point NPRS scale).

Exclusion Criteria:

* In the opinion of the Investigator, has a history of pulmonary, cardiovascular (including uncontrolled hypertension), neurologic, endocrine, hepatic, gastrointestinal, or kidney disease or therapy that, in the opinion of the Investigator, would jeopardize the patient's well being by participation in this study or is mentally or emotionally unsuitable to participate, or unable/unwilling to comply with the study assessments.
* Used opiates continuously (including tramadol) for more than ten days in the past year.
* Hypersensitivity or poor tolerance to ibuprofen or short term opioids.
* Currently receiving any medications that are not at a stable dose (the same dose for > 4 weeks prior to date of surgery).
* Was dosed with another investigational drug within 30 days prior to the Screening Visit or has previously received treatment with Q8003.
* Current therapy with central nervous system depressant medications that might increase the risks of treatment with opioids (other than those used with surgical anesthesia).
* Current evidence of alcohol abuse (regularly drinks more than 4 units of alcohol per day; 1 unit = ½ pint of beer, 1 glass of wine, or 1 ounce of spirit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2009-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Difference in pain intensity scores from baseline | 48 hours

SECONDARY OUTCOMES:
Safety: adverse events, moderate and severe reports of opioid-related adverse events | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Patricia T. Richards, MD, Ph.D., Study Director — QRxPharma Inc.
Locations (5):
- United States (5):
  - Investigator Site, Anaheim, California
  - Investigator Site, Owings Mills, Maryland
  - Investigator Site, Pasadena, Maryland
  - Investigator Site, San Antonio, Texas
  - Investigator Site, Salt Lake City, Utah